CLINICAL TRIAL: NCT06881589
Title: Ultrasound Parameters to Predict Difficult Videolaryngoscopy
Brief Title: Ultrasound Parameters for Difficult Videolaryngoscopy
Status: Recruiting | Type: Observational
Sponsor: Clinica Universidad de Navarra, Universidad de Navarra (Other)
Collaborators: County Clinical Emergency Hospital Cluj-Napoca (Other); Hospital Ancona (Unknown); Hospital CUF Porto (Unknown)
Responsible Party: Sponsor
Other Study IDs: MAFV 2
Record Dates: First submitted 2025-03-11; First posted 2025-03-18 (Actual); Last update posted 2025-03-18 (Actual); Status verified 2024-09

CONDITIONS: Difficult Videolaryngoscopy
Keywords: Ultrasound;Difficult Videolaryngoscopy

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patient undergoing general anesthesia with videolaryngoscopy intubation: Patient undergoing general anesthesia with intubation We will explore clinical airway parameters and external ultrasound parameters of the airway.
  Interventions: Diagnostic Test: Ultrasound mesurements

INTERVENTIONS:
Diagnostic Test: Ultrasound mesurements — Compare various clinical test with ultrasound parameters to predict difficult videolaryngoscopy intubation.

SUMMARY:
Ultrasound has become an essential tool for the daily work of any doctor, but in certain specialties such as Anaesthesiology, its use has greatly increased the safety offered to patients throughout the perioperative period, either to perform nerve blocks, for vascular access, intraoperative hemodynamic management or any other use that allows increasing quality of care.

DETAILED DESCRIPTION:
The management of the upper airway and the diagnosis of pathological conditions are essential skills for any doctor especially for Anaesthesiologist, ER physician, or Intensive Care physician. Because an inadequate airway management continues to be an important contributor to patient mortality and morbidity, any tool that can improve it should be considered as an addition to conventional clinical evaluation.

Unfortunately, most of the clinical parameters that should allow us to assess a potential difficult airway, do not always lead us to an adequate prediction, that is why US(Ultrasound) is use as an emerging tool in many fields, is also gathering strength in this search for a definitive predictor parameter.

Ultrasound has many obvious advantages (safe,fast, repeatable, portable, widely available and gives dynamic images in real time).

Sonographic studies are operator-dependent and although the identification of basic structures could be acquired with only a few hours of training, but more complex studies require a learning curve of months or even years. The high frequency linear probe (5-14 MHz) is probably the most suitable for the airway because images are of superficial structures (within 0-5 cm below the skin surface).

The growing academic interest in the use of US to look for predictors of difficult airway is centred mainly on measurements at the level of pretracheal tissues. But the greatest limitation of these studies is the disparity of the fat distribution that exists between different ethnic groups and and sexes, and the lack of standardization method in patient´s intubation conditions.

So, this study propose to assess different ultrasound windows at the level of pretracheal tissues such as independent predictors of Difficult Vydeolaryngoscopy.

ELIGIBILITY:
Inclusion Criteria:

* Patients (male or female) ASA I-III, aged between 18 and 90 years, undergoing scheduled surgery requiring orotracheal intubation. The signature of the informed consent is required authorizing its inclusion in the study.

Exclusion Criteria:

* Obesity class II defined as a BMI greater than 35.
* Pregnant.
* Cervical tumors, goiter or patients who have required radiotherapy at the cervical level
* Abnormalities that condition anatomy alterations such as facial / cervical fractures.
* Maxillofacial abnormalities
* People who cannot give their consent

Ages: 18 Years to 90 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Patients (male or female) ASA I-III, aged between 18 and 90 years, undergoing scheduled surgery requiring orotracheal intubation. The signature of the informed consent is required authorizing its inclusion in the study.
Sampling Method: Non-Probability Sample
Enrollment: 210 (Estimated)
Dates: Start 2023-01-27 (Actual); Primary Completion 2025-09-01 (Estimated); Study Completion 2025-09-01 (Estimated)

PRIMARY OUTCOMES:
Distance from skin to Hyoid bone measured with lineal ultrasound probe | 5 minutes
Distance from skin to epiglottis measured with lineal ultrasound probe | 5 minutes
Tongue Thickness measured with convex probe | 5 minutes
Distance from Jaw to Hyoid bone distance measured with convex probe | 5 minutes

SECONDARY OUTCOMES:
Modified Mallampati Score Class I: Soft palate, uvula, fauces, pillars visible. Class II: Soft palate, major part of uvula, fauces visible. Class III: Soft palate, base of uvula visible. Class IV: Only hard palate visible. | 1minute
Thyromental distance measured from the thyroid notch to the tip of the jaw with the head extended | 1minute
Sternomental distance the distance from the suprasternal notch to the mentum and is measured with the head fully extended on the neck and the mouth closed | 1minute
Interincisor distance DIstance in centimeters between fornt incisors | 1minute
Upper Lip Bite Test upper lip bite criteria-class I = lower incisors can bite the upper lip above the vermilion line, class II = lower incisors can bite the upper lip below the vermilion line, and class III = lower incisors cannot bite the upper lip | 1minute
neck circumference Using a flexible measuring tape in centimeters, neck circumference at the level of thethyroid cartilage will be measured | 1minute

CONTACTS AND LOCATIONS:
Locations (1):
- Clinica Universidad de Navarra, Madrid, Spain

IPD SHARING:
Plan to Share IPD: Undecided